CLINICAL TRIAL: NCT01726881
Title: Predicting Central Pain Among People With a Spinal Cord Injury by Evaluating Mechanisms Regulating Pain and Efficacy Testing of the TENS Apparatus
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: SHEBA-12-9572-GZ-SMC
Record Dates: First submitted 2012-11-08; First posted 2012-11-15 (Estimated); Last update posted 2018-08-28 (Actual); Status verified 2018-08

CONDITIONS: Pain; Healthy
Keywords: chronic; Spinal Cord Injury patients
MeSH Terms: conditions — Pain; Bronchiolitis Obliterans Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Fresh Spinal Cord Injury patients (Experimental): Spinal Cord Injury patients that are currently admitted to the rehabilitation unit with three weeks or less since injury that will over go several tests and will fill out several questionnaires.
  Interventions: Device: Thermal stimulation; Device: Mechanical stimulation
- Chronic Spinal Cord Injury patients (Experimental): Spinal Cord Injury patients with one year or more since injury that will over go several tests and will fill out several questionnaires
  Interventions: Device: Thermal stimulation; Device: Mechanical stimulation; Device: Transcutaneous Electrical Nerve Stimulator (TENS)
- Healthy volunteers (Active Comparator): Healthy subjects that will over go several tests and will fill out several questionnaires
  Interventions: Device: Thermal stimulation; Device: Mechanical stimulation

INTERVENTIONS:
Device: Thermal stimulation — Stimulation using a Thermal Sensory Analyzer:
  2001, Maddock ltd., Israel.
Device: Mechanical stimulation — Stimulation using Semmes-Weinstein-Monofilament Touch Test Sensory Evaluators
Device: Transcutaneous Electrical Nerve Stimulator (TENS) — A portable stimulator designed to Physical treatment of pain. TENS - Cedar rehab X2. Chattanooga group.USA.
  Arms: Chronic Spinal Cord Injury patients

SUMMARY:
People with a Spinal Cord Injury can develop chronic pain within months of the injury. Up to 80% of the patients will develop chronic pain called "central pain" and describe the pain as: burning, stabbing, or "like electricity." Central pain mechanism is unknown and therefore treatment is currently not effective.

It is hypothesized that chronic pain is associated with impaired function of the systems regulating pain, however, this hypothesis has not been tested among Spinal Cord Injury patients. Presence of such a connection, between the regulating system dysfunction and central pain, will help both predicting the risk of central pain and develop a treatment.

The current research objective is to make several sensory measurements which will measure the functioning mechanisms of regulation and control of the pain. These measurements are accepted throughout the world and are based on psychophysical assessment of patients. these Measurements are designed to assess whether Spinal Cord Injury chronic central pain patients demonstrate impairment in the regulation of pain. Finding such a link between central pain and impaired regulation could shed light on the mechanism of central pain. In addition, these measurements are designed to assess whether fresh spinal cord injury patients that have not yet developed central pain demonstrate impairment in the regulation of pain immediately after the injury. By repeated assessments of pain regulation capabilities, which will be made to fresh Spinal Cord Injury patients during the first months of injury, and comparing the results of these measurements between those who will develop center pain and those who will not, we could identify indicators for predicting the risk of central pain. Another goal of the study is to investigate the efficacy of central pain treatment, using a TENS, when the parameters of the TENS treatment will be built according to the level of functioning of the regulating systems of the individual.

ELIGIBILITY:
Inclusion Criteria:

* for all subjects:

  * age - 18-70
  * Cognitive status that allows voluntary cooperation understanding of instruction
* for chronic Spinal Cord Injury subjects:

  * spinal cord injury (complete and incomplete)
  * height of injury - under 7th cervical vertebra
  * time since injury - one year or more.
* for chronic Spinal Cord Injury subjects:

  * spinal cord injury (complete and incomplete)
  * height of injury - under under 7th cervical vertebra
  * time since injury - three weeks or less

Exclusion Criteria:

* subjects suffering from the following conditions: pacemaker,pregnancy,cancer, tuberculosis, thrombosis, metallic implants
* systemic diseases that affect the sensory perception (such as diabetes)
* patients with other neurological pathologies (such as head injury-TBI)
* Pregnancy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2012-12; Primary Completion 2019-08 (Estimated); Study Completion 2019-08 (Estimated)

PRIMARY OUTCOMES:
Sensitivity to thermic pain | 5 minutes
  Minimum temperature at which the patient reported pain. The subject will press a button once feeling pain. pain will be reported using a visual analog scale - a pain scale between 1-10.
Pain suppression capability | 5 minutes
  Reduction of pain in the presence of another stimulus. pain will be reported using a visual analog scale - a pain scale between 1-10.
Habituation to tonic stimulation | 5 minutes
  Gradient decrease in pain rating. pain will be reported using a visual analog scale - a pain scale between 1-10.
Temporal summation of pain | 5 minutes
  Standard rating of pain among several stimuli. pain will be reported using a visual analog scale - a pain scale between 1-10.

CONTACTS AND LOCATIONS:
Overall Officials: Gabriel Zeilig, MD, Principal Investigator — Sheba Hospital
Locations (1):
- Sheba Medical Center rehabilitaion facility, Ramat Gan, Israel